CLINICAL TRIAL: NCT07078045
Title: Oscillometric Arterial Pressure Measurements at Different Limb Sites: the CUFF-SITE Method Comparison Study
Brief Title: Oscillometric Arterial Pressure Measurements at Different Limb Sites
Acronym: CUFF-SITE
Status: Completed | Type: Observational
Sponsor: University of Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Dr. Alina Bergholz, Principal Investigator, University of Hamburg-Eppendorf
Other Study IDs: 2025-101549-BO-ff
Record Dates: First submitted 2025-07-13; First posted 2025-07-22 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Blood Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Postoperative patients with intraarterial arterial catheter
  Interventions: Other: Arterial pressure monitoring

INTERVENTIONS:
Other: Arterial pressure monitoring — We will perform oscillometric arterial pressure measurements at different limb sites.

SUMMARY:
This prospective, single-center observational study aims to evaluate the measurement performance of oscillometric arterial pressure measurements at different limb sites. Specifically, oscillometric arterial pressure measurements obtained at the upper arm, forearm, thigh, and lower leg with intraarterial arterial pressure measurements will be compared in non-cardiac surgery patients.

The results will provide insight into the reliability and accuracy of oscillometric blood pressure readings at alternative limb sites in clinical practice.

ELIGIBILITY:
Inclusion criteria:

* Consenting patients ≥18 years scheduled for elective non-cardiac surgery with general anesthesia
* Patients in whom intraarterial arterial pressure monitoring with a radial artery catheter is planned

Exclusion criteria:

* Patients with systolic arterial pressure interarm differences >20 mmHg
* Patients with severe peripheral arterial disease
* Patients with heart rhythms other than sinus rhythm
* Patients with contraindications for peripheral cuff placement (e.g., arteriovenous fistula, skin lesions)
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The CUFF-SITE study is a single-center prospective method comparison study conducted at the University Medical Center Hamburg-Eppendorf, Hamburg, Germany. A total of 84 patients scheduled for non-cardiac surgery with general anesthesia in whom intraarterial arterial pressure monitoring with a radial artery catheter is planned will be included.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2025-07-29 (Actual); Primary Completion 2025-12-15 (Actual); Study Completion 2025-12-15 (Actual)

PRIMARY OUTCOMES:
Agreement between oscillometric and intraarterial arterial pressure measurements | Immediate postoperative period, typically within a few hours after surgery (and in all cases within the first 24 postoperative hours)
  Mean ± standard deviation of the differences with 95% limits of agreement between oscillometric arterial pressure measurements obtained at the upper arm, forearm, thigh, and lower leg and intraarterial arterial pressure measurements (for mean, systolic, and diastolic arterial pressure).

SECONDARY OUTCOMES:
Correlation coefficients | Immediate postoperative period, typically within a few hours after surgery (and in all cases within the first 24 postoperative hours)
  Correlation coefficients between oscillometric arterial pressure measurements obtained at the upper arm, forearm, thigh, and lower leg and intraarterial arterial pressure measurements (for mean, systolic, and diastolic arterial pressure).
Classification of measurement differences | Immediate postoperative period, typically within a few hours after surgery (and in all cases within the first 24 postoperative hours)
  Classification of measurement differences between oscillometric arterial pressure monitoring at the upper arm, forearm, thigh, and lower leg and intraarterial arterial pressure monitoring according to their clinical relevance (for mean and systolic arterial pressure)
Percentage of oscillometric arterial pressure measurements obtained at the upper arm, forearm, thigh, and lower leg that are within ±5 mmHg of the corresponding intraarterial arterial pressure measurements | Immediate postoperative period, typically within a few hours after surgery (and in all cases within the first 24 postoperative hours)
  Percentage of oscillometric arterial pressure measurements obtained at the upper arm, forearm, thigh, and lower leg that are within ±5 mmHg of the corresponding intraarterial arterial pressure measurements (for mean, systolic, and diastolic arterial pressure)
Cross-comparisons | Immediate postoperative period, typically within a few hours after surgery (and in all cases within the first 24 postoperative hours)
  Mean ± standard deviation of the differences with 95% limits of agreement between oscillometric arterial pressure measurements obtained at the upper arm, forearm, thigh, and lower leg (for mean, systolic, and diastolic arterial pressure)

OTHER OUTCOMES:
Incidence of measurement failures | Immediate postoperative period, typically within a few hours after surgery (and in all cases within the first 24 postoperative hours)
  Incidence of measurement failures of oscillometric arterial pressure monitoring at the upper arm, forearm, thigh, and lower leg defined as any instance in which the device fails to display an arterial pressure reading or shows an error message

CONTACTS AND LOCATIONS:
Overall Officials: Alina Bergholz, MD, Principal Investigator — University Medical Centre Hamburg-Eppendorf
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany, Germany

IPD SHARING:
Plan to Share IPD: No